CLINICAL TRIAL: NCT00562874
Title: Increasing Animal Source Foods in Diets of HIV-Infected Kenyan Women and Their Children
Brief Title: Nutrition Intervention in Drug Naive HIV-infected Kenyan Women and Their Children
Acronym: HNP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University School of Health & Rehabilitation Sciences (Other)
Collaborators: United States Agency for International Development (USAID) (U.S. Federal Agency); Moi Univeristy (Other); University of California, Los Angeles (Other); Heifer Project International (Other); USDA, Western Human Nutrition Research Center (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: Indiana University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 0609-55; PCE-G-98-00036-00
Record Dates: First submitted 2007-11-21; First posted 2007-11-22 (Estimated); Last update posted 2013-04-05 (Estimated); Status verified 2013-04

CONDITIONS: HIV Infections
Keywords: HIV; AIDS; WOMEN; KENYA; NUTRITION; HIV/AIDS; treatment naive
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Meat Biscuit (Experimental): 75 women and one of their children will receive a biscuit containing dried meat as an ingredient for 5 days each week for 12 months.
  Interventions: Dietary Supplement: Meat Biscuit
- Soy Biscuit (Active Comparator): 75 women and one of their children will receive a biscuit containing soy flour as an ingredient for 5 days each week for 12 months.
  Interventions: Dietary Supplement: Soy Biscuit
- Wheat Biscuit (Sham Comparator): 75 women and one of their children will receive a biscuit containing pm;u wheat flour as a source of protein as an ingredient for 5 days each week for 12 months.
  Interventions: Dietary Supplement: Wheat Biscuit

INTERVENTIONS:
Dietary Supplement: Meat Biscuit — 75 women and one of their children will receive a biscuit containing dried meat as an ingredient for 5 days each week for 12 months. Women will receive 525 calories and 21 grams of protein per day and children will receive 350 calories and 14 grams of protein per day.
  Arms: Meat Biscuit
Dietary Supplement: Soy Biscuit — 75 women and one of their children will receive a biscuit containing soy four as an ingredient for 5 days each week for 12 months. Women will receive 525 calories and 21 grams of protein per day and children will receive 350 calories and 14 grams of protein per day.
  Arms: Soy Biscuit
Dietary Supplement: Wheat Biscuit — 75 women and one of their children will receive a biscuit containing only wheat lour as a source of protein as an ingredient for 5 days each week for 12 months. Women will receive 525 calories and 8 grams of protein per day and children will receive 350 calories and 5 grams of protein per day.
  Arms: Wheat Biscuit

SUMMARY:
Many of the 28 million people with immunodeficiency virus (HIV) and acquired immunodeficiency syndrome (AIDS) estimated to be living in sub-Saharan Africa also suffer from malnutrition. Reproductive age women, their infants and young children are among the most vulnerable for malnutrition and progression of HIV to AIDS and mortality is increased in the malnourished, as seen in Eastern and Southern Africa. The HIV Nutrition Project (HNP) research evaluates the effect of protein and micronutrients in meat on the health and nutritional well being of Kenyan women living with HIV in rural Kenya and the health and development of their children, by means of a randomized nutrition intervention. We will determine if meat in the diets of HIV- infected women and their children (1) protects the immune system and prevents severe infection, (2) prevents the loss of body mass and enhances the quality of life among drug naïve women not yet ill enough to warrant antiretroviral drugs and (3) positively impacts growth and development of vulnerable children of the HIV-infected women when compared to those given supplements with the same amount of energy but with either soya or wheat protein. The intervention food with beef protein provides significant vitamin B12, lysine and bio-available iron, zinc and selenium when compared to the soya and wheat supplements. Deficiencies of these nutrients may hasten HIV disease progression.

The findings from our project may have implications for the development of initiatives that are either sustainable or subsidized by the local, regional and/or global economies that ensure that all HIV-infected individuals have access to adequate nutrition support that includes foods that provide enough nutrients that are needed to optimize health and well-being. The knowledge gained may significantly impact other populations at high risk for decreased immune function such as those with tuberculosis and malaria.

This is a 3 arm randomized design where 225 HIV-infected rural Kenyan mothers with a CD4 between 250 and 500, WHO Stage 1 or 2, and with no co-existing infections, receive with their child, a nutrition biscuit supplement daily (5 days/week) for 12 months. These women are not yet ill enough to warrant treatment with antiretroviral drugs in Kenya and therefore a food intervention may keep them healthy longer and delay the need for drugs.

ELIGIBILITY:
HIV-infected women and their children who live in the Turbo catchment area in the Uasin Gishu District of Kenya and attend the AMPATH clinic there will be invited to participate in the study.

Inclusion Criteria:

* Women will be included if drug naïve and classified as WHO Stage 1 or 2 54 with a CD4 count greater than 250.
* The youngest child in the household between 6 months and 10 years who has no evidence of one or more OIs or illnesses will also be followed.

Exclusion Criteria:

* Women will be excluded if the initial CD4 is less than or equal to 250, they suffer from one or more OIs, are pregnant, or qualify as recipients of the AMPATH standard of care HHI, World Food Program or USAID Unimix food supplement interventions.
* Should the designated child be HIV positive with advanced disease and therefore not meet inclusion criteria, the next oldest child less than 10 years who meets the study criteria will be the designated child.

Min Age: 6 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 808 (Actual)
Dates: Start 2006-06; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
The impact of meat intake on mid-upper-arm muscle area; comparisons between groups, of changes from baseline to 3, 6, 9, 12, 15, 18 mos (intervention); 24 mos (6 mos post intervention). | 24 months

SECONDARY OUTCOMES:
The impact of meat intake on immune function (CD4 as well as percent of CD4 in the total lymphocyte); change from baseline to 6, 12, 18 mos (intervention), 24 months (6 mos post intervention)will be compared between groups | 24 months
The impact of meat intake on opportunistic infection (OI) incidence will be assessed monthly; change over time will be compared between groups from baseline through 18 mos (intervention and at 24 mos (6 mos post intervention). | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Judith A Ernst, DMSc, Principal Investigator — Indiana University
Locations (1):
- Moi University-Academic Model for the Prevention and Treatment of HIV, Eldoret, Rift Valley Province, Kenya